CLINICAL TRIAL: NCT02146404
Title: The Effect of Insulin-induced Hypoglycemia on Brain Lactate Accumulation and Regional Cerebral Blood Flow in Patients With Type 1 Diabetes Mellitus With and Without Hypoglycemia Unawareness and Non-diabetic Controls
Brief Title: The Effect of Hypoglycaemia on Brain Lactate Accumulation and Cerebral Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Diabetes Research Foundation (Other); European Foundation for the Study of Diabetes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1H_lac_acc
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia Unawareness
Keywords: Type 1 Diabetes Mellitus; Hypoglycemia unawareness; 1H MRS; Lactate
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Hig1 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Euglycemia (Active Comparator): Plasma glucose levels will be clamped at a constant value of ~5.0 mmol/l
  Interventions: Other: euglycemia
- Hypoglycemia (Experimental): Plasma glucose levels will be clamped at a stable value of ~3.0 mmol/l
  Interventions: Other: hypoglycemia

INTERVENTIONS:
Other: hypoglycemia — Blood glucose levels will be kept at ~3.0 mmol/l
  Other Names: Low blood glucose levels
  Arms: Hypoglycemia
Other: euglycemia — Blood glucose levels will be kept at ~5.0 mmol/l
  Other Names: Normal blood glucose levels
  Arms: Euglycemia

SUMMARY:
Iatrogenic hypoglycemia is the most frequent acute complication of insulin therapy in people with type 1 diabetes (T1DM). Recurrent hypoglycemic events initiate a process of habituation, characterized by suppression of hypoglycemic symptoms and lead to hypoglycemia unawareness, which in itself defines a particularly high risk of severe hypoglycemia. Recent evidence suggest a pivotal role for increased brain lactate transport capacity in the pathogenesis of hypoglycemia unawareness. However, there is uncertainty about the magnitude of this effect and whether such excess brain lactate is oxidizes as a glucose-sparing alternative energy source or acts as a metabolic regulator controlling brain glucose metabolism, oxygen consumption and cerebral blood flow.

Objective: The primary objective of this study is to investigate the effect of hypoglycemia on brain lactate accumulation and regional cerebral blood perfusion in humans. The secondary objective is to assess whether this effect is a related to hypoglycemia unawareness or a consequence of T1DM per se.

Hypothesis: The investigators hypothesize that hypoglycemia stimulates lactate transport over the blood-brain barrier leading to cerebral lactate accumulation and that this lactate accumulation is a function of prior hypoglycemic exposure frequency contributing to clinical hypoglycemia unawareness. Furthermore, the investigators expect that this effect of hypoglycemia on brain lactate accumulation is related to changes in cerebral blood flow (CBF).

ELIGIBILITY:
Inclusion criteria for healthy subjects

* Age: 18-50 years
* Body-Mass Index: 18-30 kg/m2
* Blood pressure: <160/90 mmHg

Inclusion criteria T1DM patients with normal hypoglycemic awareness

* Diabetes duration ≥ 1 year
* Age: 18-50 years
* Body-Mass Index: 18-30 kg/m2
* HbA1c: 42-75 mmol/mol (6-9%)
* Outcome Clarke questionnaire: 0-1
* Blood pressure: <160/90 mmHg

Inclusion criteria T1DM patients with hypoglycemia unawareness

* Diabetes duration ≥ 1 year
* Age: 18-50 years
* Body-Mass Index: 18-30 kg/m2
* HbA1c: 42-75 mmol/mol (6-9%)
* Outcome Clarke questionnaire: >3
* Blood pressure: <160/90 mmHg

Exclusion criteria for healthy subjects

* Inability to provide informed consent
* Presence of any medical condition that might interfere with the study protocol, such as brain injuries, epilepsy, a major cardiovascular disease event or anxiety disorders
* Use of any medication, except for oral contraceptives
* MR(I) contraindications (pregnancy, severe claustrophobia, metal parts in body)

Exclusion criteria for all T1DM patients

* Inability to provide informed consent
* Presence of any other medical condition that might interfere with the study protocol, such as brain injuries, epilepsy, a major cardiovascular disease event, anxiety disorders, or complications of T1DM (including neuropathy and retinopathy)
* Use of any other medication than insulin, except for oral contraceptives or stable thyroxine supplementation therapy
* MR(I) contraindications (pregnancy, severe claustrophobia, metal parts in body)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Brain lactate concentration | during stable euglycemia and hypoglyemia
  Concentration brain lactate measured with 1H-MRS

SECONDARY OUTCOMES:
Plasma lactate levels | during stable euglycemia and hypoglyemia
  Concentration arterial plasma lactate
Hormone response | during stable euglycemia and hypoglyemia

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan de Galan, Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud umc, Nijmegen, Netherlands

REFERENCES:
- [Background] van de Ven KC, van der Graaf M, Tack CJ, Klomp DW, Heerschap A, de Galan BE. Optimized [1-(13)C]glucose infusion protocol for 13C magnetic resonance spectroscopy at 3T of human brain glucose metabolism under euglycemic and hypoglycemic conditions. J Neurosci Methods. 2010 Jan 30;186(1):68-71. doi: 10.1016/j.jneumeth.2009.10.025. Epub 2009 Nov 11. PMID 19913052
- [Background] van de Ven KC, de Galan BE, van der Graaf M, Shestov AA, Henry PG, Tack CJ, Heerschap A. Effect of acute hypoglycemia on human cerebral glucose metabolism measured by (1)(3)C magnetic resonance spectroscopy. Diabetes. 2011 May;60(5):1467-73. doi: 10.2337/db10-1592. Epub 2011 Apr 4. PMID 21464446
- [Background] van de Ven KC, van der Graaf M, Tack CJ, Heerschap A, de Galan BE. Steady-state brain glucose concentrations during hypoglycemia in healthy humans and patients with type 1 diabetes. Diabetes. 2012 Aug;61(8):1974-7. doi: 10.2337/db11-1778. Epub 2012 Jun 11. PMID 22688331
- [Background] van de Ven KC, Tack CJ, Heerschap A, van der Graaf M, de Galan BE. Patients with type 1 diabetes exhibit altered cerebral metabolism during hypoglycemia. J Clin Invest. 2013 Feb;123(2):623-9. doi: 10.1172/JCI62742. Epub 2013 Jan 9. PMID 23298837
- [Background] Herzog RI, Jiang L, Herman P, Zhao C, Sanganahalli BG, Mason GF, Hyder F, Rothman DL, Sherwin RS, Behar KL. Lactate preserves neuronal metabolism and function following antecedent recurrent hypoglycemia. J Clin Invest. 2013 May;123(5):1988-98. doi: 10.1172/JCI65105. Epub 2013 Apr 1. PMID 23543056
- [Background] De Feyter HM, Mason GF, Shulman GI, Rothman DL, Petersen KF. Increased brain lactate concentrations without increased lactate oxidation during hypoglycemia in type 1 diabetic individuals. Diabetes. 2013 Sep;62(9):3075-80. doi: 10.2337/db13-0313. Epub 2013 May 28. PMID 23715622
- [Background] Bergersen LH, Gjedde A. Is lactate a volume transmitter of metabolic states of the brain? Front Neuroenergetics. 2012 Mar 19;4:5. doi: 10.3389/fnene.2012.00005. eCollection 2012. PMID 22457647
- [Derived] Wiegers EC, Rooijackers HM, van Asten JJA, Tack CJ, Heerschap A, de Galan BE, van der Graaf M. Elevated brain glutamate levels in type 1 diabetes: correlations with glycaemic control and age of disease onset but not with hypoglycaemia awareness status. Diabetologia. 2019 Jun;62(6):1065-1073. doi: 10.1007/s00125-019-4862-9. Epub 2019 Apr 19. PMID 31001674
- [Derived] Wiegers EC, Rooijackers HM, Tack CJ, Heerschap A, de Galan BE, van der Graaf M. Brain Lactate Concentration Falls in Response to Hypoglycemia in Patients With Type 1 Diabetes and Impaired Awareness of Hypoglycemia. Diabetes. 2016 Jun;65(6):1601-5. doi: 10.2337/db16-0068. Epub 2016 Mar 18. PMID 26993070